CLINICAL TRIAL: NCT04992286
Title: Detection, Evaluation and Monitoring of Frailties in the Elderly
Brief Title: Detection, Evaluation and Monitoring of Frailties in the Elderly (FRAGING)
Acronym: FRAGING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université d'Auvergne (Other); Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RBHP 2021 DUCLOS 2; 2021-A00367-34 (Other: ANSM)
Record Dates: First submitted 2021-06-28; First posted 2021-08-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Frailty
Keywords: Elderly; Community-dwelling; Screening; Prevention; Health
MeSH Terms: conditions — Frailty | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: all participants receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- people aged 65 years or more (Experimental): men or women, age Superior to 65 years
  Interventions: Other: questionnaire; Other: accelerometer

INTERVENTIONS:
Other: questionnaire — questionnaire to evaluate fragility
Other: accelerometer — To evaluate physical activity level

SUMMARY:
The aging of the French population is a major public health issue. Frailty is a reversible clinical state between optimal healthy aging and pathological aging. Early detection of frailty makes it possible to identify people aged 65 or over who are at risk of developing or worsen dependency and to offer them appropriate medical and/or social care adapted to their needs. The multidimensional screening program known as "ICOPE" (for "Integrated Care of Older People") promoted by the World Health Organization (WHO) aims to prevent functional decline worldwide and improve the well-being of older people. To support healthy aging, 6 intrinsic abilities are to be screened according to ICOPE: visual impairment, hearing impairment, depressive symptoms, locomotor abilities, cognitive decline and vitality. This program is intended to be developed in each country and adapted to the territories of action. The Mauriac and Vichy community health basins have a proportion of elderly people (≥60 years old) that is much higher than regional and national data, justifying the regional and national data, justifying the chosen action territories. The epidemiological characteristics of the French population and of the action territory made it possible to add to the following themes to the ICOPE recommendations: socio-economic situation, assistance to caregivers, vaccinations, drug iatrogeny, alcohol consumption, cardiovascular risk and cancer screening. The ICOPE process is organized in 5 steps: a community screening and a relay to the general practitioner to ensure a follow-up, an primary care in case of abnormality, evaluated at 3 months and then 6 months, establishment of a plan of care if necessary, possible referral to a specialist and mobilization of community resources mobilization of community resources and support for caregivers if needed.

The hypothesis is that conducting a fragility screening in a rural area (Mauriac health (Mauriac health basin) and a semi-urban area (Vichy health basin) would allow an effective would allow an effective allocation of expenses. In more detail, the costs are direct medical, direct non-medical, indirect and intangible costs, and efficiency is measured by measured by the quality of life score (LEIPAD). The hypothesis is that the early detection of people's frailties and their management improves their quality of life

DETAILED DESCRIPTION:
Prior to the frailty screening days, information letter will be sent to the people living in the territories of action in order to present them the project. The evaluation of the level of frailty will be done in 3 steps: an inclusion visit with one of the co-investigating physicians or one of the scientific collaborators. The investigating physician will verify the eligibility criteria (inclusion and non-inclusion criteria), and will propose to the person to participate in the protocol (consent). Individuals will also have the option to participate in the screening day but refuse to sign the sheet attesting to their consent, in which case none of the data concerning them will be kept and analyzed. After consent has been obtained, individuals will be instructed to participate in the questionnaire (M0), the frailty screening visit (M0), to the analysis of medical prescriptions (M0), to a debriefing visit (M0), and a follow-up telephone visit for people detected as frail (M3, M6). For 10 volunteers per screening day, a visit to present the accelerometers will also be added (M0), as well as an assessment of physical activity assessment (+7 days).

ELIGIBILITY:
Inclusion Criteria:

* Person, man or woman, aged 65 years or more, who came to attend a day dedicated to the theme organized within the CPTS of Mauriac or Vichy by medical medical, paramedical, medico-social professionals and cultural and sports and sports associations.
* Living in the Mauriac or Vichy health basin.
* Able to give informed consent to participate in the research.
* Affiliation to a Social Security system.

Exclusion Criteria:

* People who have a pathological aging defined by a chronic disease chronic disease covered by the Long Term Affection (ALD).
* Persons under guardianship or curatorship.
* Refusal to participate in the study expressed by the person.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Medico-economic relevance of early detection of frailty through a day dedicated to this theme organized in a rural and semi-urban area | Baseline
  The costs include direct medical costs (costs of screening for frailty, post-screening management, avoided by early management); direct non-medical costs (out of pockets); indirect costs (caregiver opportunity costs) measured in euros
Evaluation of precarity | Baseline
  measured by the Evaluation of Precarity and Inequalities of Health in Health Examination Centers (EPICES) score (min: 0-max: 100; lower scores referring to good conditions, 30=threshold of precarity),
Evaluation of psychological aspect | Baseline
  measured by the psychological aspect measured by the dedicated questionnaire (PHQ-9) (min: 0-max: 27; lower scores referring to good conditions),
Evaluation of quality of life | Baseline
  measured by the quality of life score (LEIPAD) (min: 0-max: 132; lower scores referring to good conditions)
Evaluation of caregiver | Baseline
  measured by the caregiver questionnaire (MiniZarit) . (min: 0-max: 7; lower scores referring to good conditions)
Medico-economic relevance of early detection of frailty through a day dedicated to this theme organized in a rural and semi-urban area (Cost effectiveness). | Baseline
  Effectiveness is measured by the quality of life score (LEIPAD) (min: 0-max: 132; lower scores referring to good conditions).

SECONDARY OUTCOMES:
Prevalence of frailty among people aged 65 or more in the Mauriac and Vichy community health regions. | Baseline
  measured in pourcent (%)
Prevalence of vaccination rate among people aged 65 or more in the Mauriac and Vichy community health regions. | Baseline
  measured in pourcent (%)
Prevalence of the rate of organized cancer screening among people aged 65 or more in the Mauriac and Vichy community health regions. | Baseline
  measured in pourcent (%)
Prevalence of the rate of risky alcohol consumption among people aged 65 or more in the Mauriac and Vichy community health regions. | Baseline
  measured in pourcent (%)
Prevalence of participants with a high cardiovascular risk factor among people aged 65 or more in the Mauriac and Vichy community health regions. | Baseline
  measured in pourcent (%)
Identify the determinants of frailty (physical, psychological, and associated factors) in people aged 65 years or more in a rural and a semi-urban population. | Baseline
  measured by physical examination by physician
To measure physical activity levels of 65 years or older in a rural and a semi-urban population | Baseline
  measured by the questionnaire (ONAPS-Q) and by accelerometer (MET.minutes/week)
To measure physical inactivity levels of 65 years or older in a rural and a semi-urban population | Baseline
  measured by - sedentary time measured by the questionnaire (ONAPS-Q) and by accelerometer (minutes per day) (no scale)
Modeling the flow of screened and identified frail participants who will be managed by type of frailty identified | Baseline
  - Categorization of the health pathways followed by the study cohort (no unit of measure)
Modeling the flow of screened and identified frail participants who will be managed by type of frailty identified (monte Carlo microstimulation) | Baseline
  measured by - Monte Carlo micro-simulation that will model the flows of participants (no unit of measure)

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France